CLINICAL TRIAL: NCT00275652
Title: A Randomized, Double-Blind Trial of Telbivudine (LdT) Versus Lamivudine in Adults With Decompensated Chronic Hepatitis B and Evidence of Cirrhosis.
Brief Title: A Comparison of the Drug Telbivudine (LdT) and Lamivudine in Adults With Decompensated Chronic Hepatitis B and Evidence of Cirrhosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207-04
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Hepatitis B; Cirrhosis
MeSH Terms: conditions — Hepatitis B; Fibrosis | interventions — Telbivudine; Lamivudine

INTERVENTIONS:
Drug: LdT (Telbivudine) and lamivudine

SUMMARY:
This trial is being done to see if the investigational drug, LdT (Telbivudine), is safe and effective in the treatment of hepatitis B infection. In addition to this, we will be looking at the comparison of the effects (good and bad) of LdT and lamivudine.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded trial looking at the drug Telbivudine (LdT) and comparing it to the drug lamivudine in patients with chronic hepatitis B and evidence of Cirrhosis.

Interested participants will first be seen for a screening visit, to determine eligibility for the study. Participants will have a medical history taken along with a physical exam and a blood draw. Prior to receiving the study drug, participants may be required to have a liver biopsy. If one was done in the past 5 years, it may be possible to use the results of the previous biopsy. If participants are unable to have a liver biopsy due to medical reasons, an ultrasound, CT, or MRI scan may be done instead. If an imaging study has been done in the past two years, it may be possible to use the results from this test.

All eligible participants will be put into one of two groups by chance (as in the flip of a coin). One group will receive 600 mg of LdT (3 tablets) plus a lamivudine placebo capsule (1 sugar pill) daily. While the other group will be receiving 100 mg of lamivudine (1 capsule) plus 3 LdT tablets (3 sugar pills) daily. Participants will take the study drug daily for a total of 104 weeks (2 years).

Participants will return for clinic visits at weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 52, 60, 68, 76, 84, 92, 100, and 104. Participant's vital signs (temperature, pulse, weight) and blood samples will be collected at each visit.

If after one year of being on the drug, there is no hepatitis b found in your blood, you may be stopped from the study drug. Participants will continue to be required to return to the clinic for study visits so information can be continued to be collected and for your condition to be monitored. If future blood tests show that the hepatitis B virus returned, participants will be told to restart their study drug.

At the end of the 104 weeks or if the treatment was stopped early for any reason except a liver transplant, or if additional treatment was not chosen for hepatitis B, participants will be asked to return to the clinic once every four weeks for 4 months. For each return visit to the clinic, vital signs and blood samples will be collected and recorded. A physical exam will be at the last follow-up visit.

If the study was stopped due to a liver transplant, participants will be asked to return for clinic visits at 4 and 16 weeks after surgery. At these visits, no procedures will be done, but a review of the participant's medical record.

Participants will be involved for 2 years and 4 months.

ELIGIBILITY:
Patients with chronic hepatitis b with evidence of cirrhosis, who are at least 18 to 70 years old, may be eligible to participate in this study.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2004-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
A composite endpoint called "clinical response" which is defined as HBV DNA <10 4 copies/ml and normal ALT and improvement, or stabilization in CTP score.
Durability of clinical response
Proportion of patients achieving improvement, stabilization, and worsening in CTP score
Proportion of patients with normal ALT
Improvements in serum albumin levels, in patients with hypoalbuminemia pre-treatment

SECONDARY OUTCOMES:
Time to clinical response
Duration of clinical response
Proportion of patients achieving improvement, stabilization, and worsening in CTP score
Improvement, stabilization, and worsening in a modified CTP score.
ALT normalization.

CONTACTS AND LOCATIONS:
Overall Officials: W. Ray Kim, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States